CLINICAL TRIAL: NCT03665740
Title: A Pilot RCT on the Effect of Resveratrol on Mood, Memory Deficits, Hippocampal Inflammation and Neurogenesis in Veterans With Gulf War Illness
Brief Title: Multimodal Investigation of the Neuroprotective Effects of Resveratrol (MINER)
Acronym: MINER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VISN 17 Center of Excellence (U.S. Federal Agency)
Collaborators: Texas A&M University (Other); Baylor University (Other); KR Love Quantitative Consulting and Collaboration (Other)
Responsible Party: Principal Investigator, Dena Davidson, Director of Research, VISN 17 Center of Excellence
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW160050
Record Dates: First submitted 2018-08-08; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Gulf War Illness
Keywords: Gulf War Illness; Chronic Multisymptom Illness; Antioxidants; Resveratrol; Gulf War Syndrome
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: Randomized Double-blind Placebo controlled, intent-to-treat
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Experimental): Doses of resveratrol at 500 mg will begin with a dose titration period. In order to reach a maximum dose of 2000 mg for the resveratrol, titration will begin at 500 mg for 6 weeks, then increased to 1000 mg for 6 weeks and increased to 1500 mg for 6 weeks and increased to 2000 mg for the remaining 6 weeks on treatment.
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator): Doses of placebo at 500 mg will begin with a dose titration period. In order to reach a maximum dose of 2000 mg for the placebo, titration will begin at 500 mg for 6 weeks, then increased to 1000 mg for 6 weeks and increased to 1500 mg for 6 weeks and increased to 2000 mg for the remaining 6 weeks on treatment
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Resveratrol — resveratrol is an OTC supplement

SUMMARY:
Since their return from military service in the 1990-1991 Gulf War, many Veterans have been affected by debilitating symptoms that are not easily explained. A leading hypothesis states that the combination of exposure to toxic chemicals and environmental stressors are responsible for a cluster of debilitating symptoms known as Gulf War Illness (GWI). Research has found that over-the-counter antioxidant supplements such as resveratrol may reverse the damage that causes these debilitating symptoms. Resveratrol is a nutrient found abundantly in the skin of red grapes that is known to have robust antioxidant and anti-inflammatory properties. The investigators predict that resveratrol treatment will improve memory issues, difficulties with thinking and mood problems in Veterans with GWI and that resveratrol will do so with minimal risk.

DETAILED DESCRIPTION:
A randomized controlled trial is proposed that will employ well-validated instruments and state-of-the-art techniques to assess improvements in cognitive functioning, functional status, mood, hippocampal neurogenesis and functional connectivity as well as anti-inflammatory and antioxidant effects of treatment with resveratrol. Design: The proposed study will be an intent-to-treat outpatient, randomized, double-blind, clinical trial of 93 Veterans who meet the Centers for Disease Control and Prevention and Kansas case definitions for GWI.

The study involves a comparison of resveratrol at a dose of 2000 mg and placebo. All doses will be administered orally once or twice daily. Doses of resveratrol at 500 mg will begin with a dose titration period. In order to reach a maximum dose of 2000 mg for the resveratrol, titration will begin at 500 mg for 6 weeks, then increased to 1000 mg for 6 weeks and increased to 1500 mg for 6 weeks and increased to 2000 mg for the remaining 6 weeks on treatment. Morning dosing will be taken with or before breakfast. Evening dosing will be taken with or before dinner.

ELIGIBILITY:
Inclusion Criteria:

1. Served on active military duty and deployed to the Persian Gulf region August 1990 - July 1991;
2. English speaking and able to understand the consent form and study questionnaires;
3. Willing and able to be randomized to treatment and to commit to a 26-week study;
4. Men and women between the ages of 44 to 68 (the number of 1990-1991 Gulf War Veterans who are older than 68 dramatically decreases because many of those with GWI have died prematurely);
5. Meet the Kansas case definition for the diagnosis of GWI as well as the more inclusive CDC definition
6. Stabilization on any psychiatric medication (≥3 months on selective serotonin reuptake inhibitor or monoamine oxidase inhibitor, ≥1 month on anxiolytic or beta-blockers);
7. Female subjects of childbearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test and agree to use reliable method of birth control (for example, oral contraceptives or Norplant; a reliable barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam]; intrauterine devices; partner with vasectomy; or abstinence) during the study. Note that this inclusion criterion applies only to females of childbearing potential. Females of childbearing potential are defined as women not surgically sterilized and between menarche and 2 years post-menopause.

Exclusion Criteria:

1. Unstable or poorly controlled diabetes type II (HbA1C >9.0);
2. Cancer;
3. Lifetime diagnosis of schizophrenia or bipolar disorder or a history of psychiatric hospitalization for, or current diagnosis (i.e., the past 6 months) of substance dependence;
4. Major depressive disorder or posttraumatic stress disorder requiring hospitalization;
5. Significant CNS disease including TIAs or stroke, dementia, syncopal episodes, severe head trauma, multiple sclerosis;
6. Serious or advanced heart disease or clinically relevant abnormal electrocardiogram (ECG) or postural hypotension;
7. Untreated sleep apnea or body mass index (BMI) placing patients at risk for undiagnosed sleep apnea (BMI≥35 kg/m2);
8. Subjects with renal insufficiency or chronic renal disease defined by national Kidney Foundation Disease Outcome Quality Initiative criteria (2000) with a GFR less than or equal to 90 mL/min/1.73m2. Laboratory monitoring of CR and Bun and eGFR will be obtained at baseline and prior to each titration and at study end or early termination. If Cr and Bun increase above upper limit of normal and eGFR drops to <45 or more than 35% the study drug will be discontinued and a nephrology consult will be ordered;
9. Liver enzymes >3 times normal on 3 consecutive laboratory tests; evidence of significant hepatocellular injury as evidenced by elevated serum levels of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 3 times the upper limit of normal (ULN); total or indirect bilirubin greater than 1.2 x ULN; alkaline phosphatase greater than 1.5 x ULN; prothrombin time (PT) as INR greater than 2.4 x ULN; or albumin less than 1 times the lower limit of normal (LLN) at baseline. Resveratrol is only anticipated to affect LFTs indirectly, by slowing statin metabolism. Persistent significant elevation of amino transferases are defined as >3x normal of normal upper limit on 2 consecutive measurements. Under the conditions of high dose statin therapy, it is typically addressed by temporarily stopping statin administration, then slowly titrating the dose back up under careful observation. Failure to reduce aminotransferase levels after the temporary cessation of statins (and a third LFT measurement is taken) would necessitate cessation of resveratrol treatment.
10. Use of cytochrome P450 3A4 substrates with high risk of toxicity (e.g., terfenadine, cisapride, astemizole, disopyramide, amiodarone, dronedarone, colchicine, cyclosporine, quinidine, pimozide, cisapride, amlodipine, felodipine, nicardipine, nifedipine, nisoldipine, nitrendipin, nimodipine and verapamil);
11. Use of blood thinners (e.g., Coumadin);
12. Use of resveratrol-containing supplements.

    Participation in the scanning portion of the study is not required to participate in the clinical trial. Subjects who are interested in the scanning study will be asked to sign a second consent and will be screened for MRI-specific exclusion criteria. The additional exclusion criteria for participating in the MRI portion are listed below.
13. General medical conditions that would prevent the participant from completing MRI scanning (active seizure disorder, dementia, active back or muscle spasms);
14. Positive MRI safety screen for metal or history of penetrating head or eye wound without subsequent radiological evidence that the wound is metal-free;
15. Participants that are (were) welders or that have had metal surgically removed from their eyes without radiological evidence that the wound is metal-free;
16. MRI quality problems (tremors, significant claustrophobia);
17. Shrapnel or other metal embedded in the body;
18. Implanted orthopedic devices (e.g., metal rods, plates or screws but excluding nonferrous material);
19. Implanted metal devices or prosthetics, or mechanical implants (e.g., pacemakers, electrical implants, cochlear implants);
20. Implanted contraceptive devices (excluding those made of nonferrous material);
21. Outside devices made of metal (e.g., neck braces, surgical staples, or artificial limbs), or non-removable dentures, braces or other metal orthodontics;
22. Tattoos not done professionally or non-removable body piercings.

Ages: 44 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Cognitive Function | Baseline & Post (week 26)
  CVLT-II: measure of cognitive functioning and memory
Change from baseline in Mood | Baseline, Mid (week 13) and Post (week 26)
  Beck Depression Inventory II
Change from baseline in Daily Functioning | Baseline and Post (week 26)
  WHODAS 2.0: measure of disability and global health

SECONDARY OUTCOMES:
Change from baseline in Structural MRI Scans | Baseline & Post (Week 26)
  Structural MRI scanning of hippocampus
Change from baseline in Diffusion Tensor Imaging | Baseline & Post (Week 26)
  A diffusion tensor imaging scan of hippocampus

OTHER OUTCOMES:
Change from baseline in Pro-inflammatory cytokines | Baseline & Post (Week 26)
  IL-1β; TNF-α; IL-6; IL-1α; Interferon-Y; G-CSF/CSF3; GM_CSF/CSF2; IL-8; IP-10; RANTES; Resistin; PAI-1; IL-12; IL-13; Eotaxin-3; MCP-1; MIP-1α; IL-2; Leptin; Adiponectin; IL-17α; IL-4; IL10

CONTACTS AND LOCATIONS:
Overall Officials: Dena Davidson, Ph.D., Principal Investigator — VISN 17 Center of Excellence
Locations (1):
- VISN 17 Center of Excellence for Research on Returning War Veterans, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for the VISN 17 Center of Excellence for Research on Returning War Veterans — https://www.mirecc.va.gov/visn17